CLINICAL TRIAL: NCT05754099
Title: Identification of Clinically Significant Markers of Hereditary Transthyretin Amyloidosis (TTR) in Pre-symptomatic Mutation Carriers: a Prospective Longitudinal Multicentre Study
Brief Title: Identification of Clinically Significant Markers of ATTRv in Pre-symptomatic Mutation Carriers.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4108
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-02

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this prospective observational study is to periodically monitor pre-symptomatic subjects carrying a mutation of Transthyretin (TTR), identified in the context of a family screening of affected proband, through instrumental methods and clinical scales in order to identify the first signs of clinically significant organ involvement by the disease. Healthy asymptomatic carriers will be subjected to regular monitoring through clinical evaluations and instrumental investigations defined by the consensus group (Conceicao et al.) in order to validate the criteria defined by this group to define the onset of the disease. A subgroup of carriers with scales and instrumental tests negative for damage to the peripheral nervous system or cardiac, but with subjective symptoms compatible with the disease, will be subjected to further instrumental tests not indicated by consent.

ELIGIBILITY:
Inclusion criteria

1. Pre-symptomatic carriers of TTR mutation in regular follow-up at the Centres.
2. Signature of the written informed consent.
3. Age not less than 10 years compared to the age of onset of the relative with the youngest age of onset and/or a history of bilateral carpal tunnel syndrome undergoing surgery.

Exclusion criteria

* Other causes of neuropathies (diabetes; MGUS; alcoholism; vitamin deficiency).
* Other causes of hypertrophic heart disease.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Data from pre-symptomatic carriers who have signed the written informed consent, in regular follow-up at the Centres, will be included in the study. Carriers recruited should be no less than 10 years of age compared to the age of onset of the affected relative with the youngest age of onset or should have a history of bilateral carpal tunnel syndrome undergoing surgery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of a cohort of pre-symptomatic subjects carrying a TTR mutation | 3 years
  To evaluate in a cohort of pre-symptomatic subjects carrying a TTR mutation the disease onset according to the European consensus criteria (Conceicao et al.).

CONTACTS AND LOCATIONS:
Locations (1):
- Flavia Torlizzi, Roma, Italy